CLINICAL TRIAL: NCT02124837
Title: An Intervention Study to Investigate the Effect of Different Types of Break Activities on Workers´ Psychological and Physiological Health & Job Performance
Brief Title: Intervention Study on Break Activities and Workers´ Psychological and Physiological Health & Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Jessica de Bloom, Dr., Tampere University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 257682SA
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Exposure to Nature During Lunch Breaks; Relaxation Exercises During Lunch Breaks
Keywords: lunch breaks, recovery, nature, park walking, relaxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Participants continue their normal lunch routine.
- Relaxation exercise during lunch break (Experimental): Participants perform relaxation exercises during each lunch break during work for a period of 2 working weeks.
  Interventions: Behavioral: Relaxation during lunch break
- Park walk during lunch break (Experimental): Participants go for a walk in the closest park nearby each lunch break during work for a period of 2 working weeks.
  Interventions: Behavioral: Park walk during lunch break

INTERVENTIONS:
Behavioral: Park walk during lunch break
  Arms: Park walk during lunch break
Behavioral: Relaxation during lunch break
  Arms: Relaxation exercise during lunch break

SUMMARY:
The objective of this research project is to understand and to improve workers´ recovery from work stress. Although recovery during lunch breaks is the most common within-workday break, it has received only minor research attention. Therefore, we will study whether lunch breaks including a relaxation session or exposure to nature have more favorable outcomes than usually spent lunch breaks concerning: a) recovery processes, b) health, c) well-being, d) job performance and e) creativity. We approach recovery by combining the theoretical frameworks of work and environmental psychology.

DETAILED DESCRIPTION:
We conduct an intervention study in a sample of 200 knowledge-workers who engage in different lunch break activities for 15-minutes per day, two weeks in a row. We randomly assign participants to three experimental conditions: 1) exposure to nature, 2) relaxation and 3) control group (lunch break spent as usual). Online questionnaires before and after the intervention assess long term changes regarding recovery processes and the major outcome variables. Before, during and after the intervention, SMS and paper-pencil questionnaires measure the same constructs four times a day with fewer items. We also measure blood pressure and collect saliva samples to map cortisol excretion across the intervention period. A timed experimental task (i.e., the Alternative Uses Task) is used to examine differences in creativity between the three groups after the intervention period.

By combining the knowledge of work and environmental psychology about recovery and restorative experiences, by merging three recovery perspectives (settings, processes, and outcomes) and by using data triangulation, we produce valid results that broaden our view on mechanisms underlying recovery and enhance our understanding about their links to psychological, behavioural and physiological outcomes, resulting in a more comprehensive picture of work stress recovery in general.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Finnish language
* Paid work for at least 24 hours per week

Exclusion Criteria:

* Shift work, highly irregular working hours
* Serious illness or allergies that prevent participants from walking in nature

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Well-being | 7 weeks
  Questionnaire data
Job performance | 7 weeks
  Questionnaire data
Creativity | 7 weeks
  Questionnaire data
Health | 7 weeks
  Questionnaire data
Salivary cortisol | 7 weeks
  Collection of saliva samples, 3 times per day, 2 times a week for a period of 7 weeks
Blood pressure | 7 weeks
  Self-administered blood pressure measurements, 3 times per day, 2 days per week for a period of 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Kinnunen, Prof., Principal Investigator — Tampere University; Kalevi Korpela, Prof., Principal Investigator — Tampere University
Locations (1):
- University of Tampere, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] de Bloom J, Kinnunen U, Korpela K. Exposure to nature versus relaxation during lunch breaks and recovery from work: development and design of an intervention study to improve workers' health, well-being, work performance and creativity. BMC Public Health. 2014 May 22;14:488. doi: 10.1186/1471-2458-14-488. PMID 24885178